CLINICAL TRIAL: NCT06816641
Title: Surgical Evacuation Of Spontaneous Intracerebral Hematoma: Clinical Outcomes and Prognostic Factors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed AHmed Ragheb, Demonstrator of Neurosurgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-1-06MS
Record Dates: First submitted 2025-01-30; First posted 2025-02-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Intracerebral Haemorrhage (ICH)
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical evacuation of Intracerebral hemorrhage (Other): Surgical evacuation of Intracerebral hematoma
  Interventions: Procedure: Surgical Evacuation of Intracerebral Hemorrhage

INTERVENTIONS:
Procedure: Surgical Evacuation of Intracerebral Hemorrhage — Surgical Evacuation of Intracerebral Hemorrhage

SUMMARY:
The aim of this study is to assess the safety and efficacy of surgical evacuation of spontaneous intracerebral hemorrhage.

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage (ICH), i.e., nontraumatic hemorrhage into the brain parenchyma with or without ventricles, is a severe type of stroke with high mortality rates. Systemic arterial hypertension and cerebral amyloid angiopathy represent the two main risk factors of primary ICH. (1) ICH is understood to injure surrounding brain tissue through the direct pressure effects of an acutely expanding mass lesion and through secondary physiological and cellular pathways triggered by the hematoma and its metabolized blood products. Direct pressure effects can include both local compression of immediately surrounding brain tissue and more widespread mechanical injury caused by increased intracranial pressure (ICP), hydrocephalus, or herniation. Early hematoma expansion, possibly driven by mechanical shearing of surrounding vessels by the initial hematoma, is common and a consistent predictor of worse ICH outcome. Secondary physiological and cellular injury mechanisms postulated to be triggered by ICH include cerebral edema, inflammation, and biochemical toxicity of blood products such as hemoglobin, iron, and thrombin. Several of the major medical therapies for ICH such as BP lowering and reversal of anticoagulation are aimed at limiting hematoma expansion. The search for effective medical treatments for protecting tissue from secondary post-ICH injury, like the search for effective neuroprotectants for ischemic stroke, has to date been unsuccessful. Surgical hematoma evacuation through craniotomy or minimally invasive approaches is aimed at both preventing further pressure-related injury and protecting against secondary physiological and cellular injury. (2) Hematoma evacuation may have therapeutic potential, based on the theoretical advantages of preventing or correcting the acute effects of hematoma and its blood products into the surrounding healthy brain parenchyma. However, because the most common sites of spontaneous ICH are the deep brain structures, such as the basal ganglia and the thalamus, a large layer of healthy brain tissue would be damaged. Additionally, neurosurgical procedures are not free of risks and adverse effects. Post-surgical complications (e.g., hemorrhages and infections) are common in this clinical scenario and carry high rates of morbidity and mortality. (3) Recent meta-analyses suggested the benefits of neurosurgical hematoma evacuation, especially when performed earlier and done using minimally invasive procedures. In MISTIE III (Minimally invasive surgery plus alteplase for intracranial hematoma evacuation), to confirm hemostasis and reduce the risk of rebleeding, the mean time from onset of ICH to surgery was 47 hours while the mean time from onset of ICH to treatment completion was 123 hours. Theoretically, the earlier the hematoma is removed, the better the outcome. Therefore, a higher rate of hematoma reduction within an earlier time course may be beneficial. (4) Although the role of open surgery to treat patients with spontaneous ICH remains controversial, the use of craniotomy for intracerebral hematoma drainage is the most common strategy applied in most centers and also the most studied approach so far. (5) Controversy remains over the efficacy of surgery for ICH, particularly in the early (<12 hours) and very early (<8 hours) time windows. Further data are needed before definitive conclusions can be reached. However, the sum of preclinical and clinical data strongly suggests that early evacuation may be a necessary component of any successful surgical approach. Furthermore, recent data have suggested improved safety of such procedures using modern minimally invasive approaches. Such approaches may minimize collateral injury, allow safe management of intraoperative bleeding, and prevent postoperative rebleeding, all of which may facilitate the potential value of early ICH evacuation. (6)

ELIGIBILITY:
Inclusion Criteria:

* • Patients with radiological findings of ICH.

  * Age group 20-70 years.

Exclusion Criteria:

* • Traumatic ICH or ruptured aneurysm or AVM or brain tumor.

  * Postoperative cranial surgery ICH.
  * Secondary hydrocephalus.
  * Patients with other comorbidities e.g., Liver cell failure and renal cell failure.
  * Patients with bleeding disorders.
  * Patients who are regular on anticoagulant or antiplatelet therapy.
  * Small sized ICH< 30 ml.
  * GCS less than 6 preoperatively.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Morbidity after surgical evacuation of Intracerebral hematoma | 1 month
  Complications within first month
Mortality after surgical evacuation of Intracerebral hematoma | 1 month
  Death of patient within first month

SECONDARY OUTCOMES:
Morbidity after surgical evacuation of Intracerebral hematoma | 3 months
  Complications from end of 1st month to end of 3rd month
Mortality after surgical evacuation of Intracerebral hematoma | 3 months
  Death of patient

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Asch CJ, Luitse MJ, Rinkel GJ, van der Tweel I, Algra A, Klijn CJ. Incidence, case fatality, and functional outcome of intracerebral haemorrhage over time, according to age, sex, and ethnic origin: a systematic review and meta-analysis. Lancet Neurol. 2010 Feb;9(2):167-76. doi: 10.1016/S1474-4422(09)70340-0. Epub 2010 Jan 5. PMID 20056489
- [Background] Wilkinson DA, Pandey AS, Thompson BG, Keep RF, Hua Y, Xi G. Injury mechanisms in acute intracerebral hemorrhage. Neuropharmacology. 2018 May 15;134(Pt B):240-248. doi: 10.1016/j.neuropharm.2017.09.033. Epub 2017 Sep 22. PMID 28947377
- [Background] Wong JM, Ziewacz JE, Ho AL, Panchmatia JR, Kim AH, Bader AM, Thompson BG, Du R, Gawande AA. Patterns in neurosurgical adverse events: open cerebrovascular neurosurgery. Neurosurg Focus. 2012 Nov;33(5):E15. doi: 10.3171/2012.7.FOCUS12181. PMID 23116095